CLINICAL TRIAL: NCT03981744
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Ustekinumab in Participants With Active Polymyositis and Dermatomyositis Who Have Not Adequately Responded to One or More Standard-of-care Treatments
Brief Title: A Study of Ustekinumab in Participants With Active Polymyositis and Dermatomyositis Who Have Not Adequately Responded to One or More Standard-of-care Treatments
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study did not meet the primary endpoint.
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108618; CNTO1275DMY3001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Results first posted 2024-05-13 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Polymyositis; Dermatomyositis
MeSH Terms: conditions — Polymyositis; Dermatomyositis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Ustekinumab (Experimental): Participants will receive body weight-range based IV dosing of approximately 6 milligram per kilogram (mg/kg) of ustekinumab at Week 0 followed by ustekinumab 90 milligram (mg) subcutaneously (SC) at Week 8 and every 8 Weeks (q8w) administrations through Week 72. At Week 24, participants will receive IV dosing of placebo.
  Interventions: Drug: Ustekinumab 6 mg/kg; Drug: Ustekinumab 90 mg; Drug: Placebo IV
- Group 2: Placebo (Placebo Comparator): Participants will receive IV dosing of placebo at Week 0 followed by placebo SC administrations at Weeks 8,16 and 24. At Week 24, participants will receive body weight-range based IV dosing of approximately 6 mg/kg of ustekinumab, followed by ustekinumab 90 mg SC q8w administrations Week 32 through Week 72.
  Interventions: Drug: Ustekinumab 6 mg/kg; Drug: Ustekinumab 90 mg; Drug: Placebo IV; Drug: Placebo SC

INTERVENTIONS:
Drug: Ustekinumab 6 mg/kg — Participants will receive body weight-range based IV dosing of 6 mg/kg of ustekinumab at Week 0 in Group 1 and at Week 24 in Group 2.
  Other Names: STELARA
Drug: Ustekinumab 90 mg — Participants will receive ustekinumab 90 mg SC at Week 8 and every 8 Weeks (q8w) through Week 72 in Group 1 and q8w Week 32 through Week 72 in Group 2.
  Other Names: STELARA
Drug: Placebo IV — Participants will receive IV dosing of placebo at Week 24 in Group 1 and at Week 0 in Group 2.
Drug: Placebo SC — Participants will receive SC dosing of placebo at Weeks 8,16 and 24.
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of ustekinumab in participants with active polymyositis (PM)/dermatomyositis (DM) despite receiving 1 or more standard-of-care treatments (for example, glucocorticoids and/or immunomodulators).

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of polymyositis (PM)/ dermatomyositis (DM) made or confirmed by a physician (such as a rheumatologist, neurologist, or dermatologist) experienced in treatment of PM/DM at least 6 weeks prior to first dose of the study drug
* Has PM or DM which is considered active despite receiving at least 1 standard-of-care treatment by the investigator
* Must be receiving 1 or more of the following protocol-permitted, systemic standard-of-care treatments: i) glucocorticoids, ii) 1 or 2 of the following immunomodulatory drugs: mycophenolate mofetil, azathioprine, oral methotrexate, oral tacrolimus, or oral cyclosporine A
* Regular or as needed treatment with topical use of glucocorticoids are permitted to treat skin lesions on a stable dose for greater than or equal to (>=) 2 weeks prior to first dose of the study drug
* Contraceptive (birth control) use by men or women should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies
* Must be medically stable on the basis of clinical laboratory tests performed at screening. If the results of the clinical laboratory tests are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant
* Demonstrable muscle weakness at screening and Week 0 measured by the Manual Muscle Testing (MMT)-8 less than or equal to (<=)135 units
* Demonstrable muscle weakness at screening measured by any 2 or more of the followings: (i) PhGA greater than or equal to (>=) 1.5 centimeter (cm), (ii) 1 or more muscle enzymes (Creatine kinase [CK], and aldolase) >=1.4*upper limit of normal (ULN), (iii) Myositis disease activity assessment tool (MDAAT)-Extramuscular Global Assessment >=1.5 cm

Exclusion Criteria:

* Has myositis other than PM/DM, including but not limited to amyopathic dermatomyositis (ADM), clinically amyopathic DM, juvenile DM, inclusion body myositis (IBM) immune-mediated necrotizing myopathy diagnosed based on muscle biopsy findings and positive anti-SRP or anti-HMGCR antibody, drug-induced myositis, PM associated with human immunodeficiency virus (HIV), and muscular dystrophy, congenital myopathy, metabolic myopathy, and mitochondrial myopathy
* Has other inflammatory diseases that might confound the evaluations of efficacy, including but not limited to rheumatoid arthritis (RA), psoriatic arthritis (PsA), systemic lupus erythematosus (SLE), psoriasis, or Crohn's disease
* Has severe respiratory muscle weakness confirmed by the investigator based on the consultation with a pulmonologist and the measures of respiratory muscle strength such as maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) and/or maximal voluntary ventilation (MVV) measurements and lung capacity such as forced vital capacity (FVC). The results need to be within population appropriate normal limits
* Has severe muscle damage (Myositis Damage Index-VAS [Muscle Damage] greater than (>) 7 centimeter [cm]), permanent weakness due to a non-IIM cause, or myositis with cardiac dysfunction
* Has glucocorticoid-induced myopathy which the investigator considers the primary cause of muscle weakness
* Has positive test result of anti-melanoma differentiation-associated protein 5 (MDA5) antibody (anti clinically amyopathic dermatomyositis (C-ADM)-140 antibody).
* Has had a nontuberculous mycobacterial infection or opportunistic infection
* Has a history of, or ongoing, chronic or recurrent infectious disease
* Has past history of severe Interstitial lung disease (ILD) flare, severe non-infectious lung inflammation which required active intervention, or multiple relapses of these conditions
* Presence or history of malignancy within 5 years before screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (32):
- Japan (32):
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Fukushima Medical University Hospital, Fukushima
  - Shinko Hospital, Hyōgo
  - Tokai University Hospital, Isehara
  - Kagoshima University Hospital, Kagoshima
  - St Marianna University Hospital, Kanagawa
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano
  - Hospital of the University of Occupational and Enviromental Health, Kitakyushu
  - Kumamoto University Hospital, Kumamoto
  - Kurashiki Central Hospital, Kurashiki
  - Shinshu University Hospital, Matsumoto
  - Minaminagano Medical Center Shinonoi General Hospital, Nagano
  - Nagasaki University Hospital, Nagasaki
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Niigata University Medical And Dental Hospital, Niigata
  - Okayama City General Medical Center Okayama City Hospital, Okayama
  - Saga University Hospital, Saga
  - Kitasato University Hospital, Sagamihara
  - Sakai City Medical Center, Sakai
  - Tohoku University Hospital, Sendai
  - Tohoku Medical And Pharmaceutical University Hospital, Sendai
  - Dokkyo Medical University Hospital, Shimotsuga Gun
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku Ku
  - The Jikei University Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
  - Ehime University Hospital, Tōon
  - University of Tsukuba Hospital, Tsukuba
  - Yamaguchi University Hospital, Ube
  - Yokohama Rosai Hospital, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Kawahata K, Ishii T, Gono T, Tsuchiya Y, Ohashi H, Yoshizawa K, Zheng R, Ayabe M, Nishikawa K. Phase 3, multicentre, randomised, double-blind, placebo-controlled, parallel-group study of ustekinumab in Japanese patients with active polymyositis and dermatomyositis who have not adequately responded to one or more standard-of-care treatments. RMD Open. 2023 Aug;9(3):e003268. doi: 10.1136/rmdopen-2023-003268. PMID 37652554

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo (matching to ustekinumab) intravenously (IV) at Week 0, then placebo subcutaneously (SC) every 8 weeks (q8w) at Weeks 8 and 16.
- Ustekinumab: Participants received body weight-range based IV dose of ustekinumab 6 mg/kg at Week 0 followed by ustekinumab 90 mg as SC injection at Weeks 8 and 16.
- Placebo to Ustekinumab: Participants who received placebo (matching to ustekinumab) intravenously (IV) at Week 0, placebo subcutaneously (SC) every 8 weeks (q8w) at Weeks 8 and 16, then in order to gain benefit from this study participants received body weight-range based IV dose of ustekinumab 6 milligrams per kilograms (mg/kg) and placebo SC (to maintain blinding) at Week 24, followed by ustekinumab 90 milligrams (mg) SC q8w thereafter through Week 72.
- Ustekinumab Through End of Study (EOS): Participants who received body weight-range based IV dose of ustekinumab 6 mg/kg at Week 0, ustekinumab 90 mg as SC injection at Weeks 8 and 16 then received placebo IV (to maintain blinding) and ustekinumab 90 mg SC at Week 24 and ustekinumab 90 mg SC q8w thereafter through Week 72.
Period: First Intervention (Prior to Week 24)
Arm/Group | Placebo | Ustekinumab | Placebo to Ustekinumab | Ustekinumab Through End of Study (EOS)
Started | 26 | 25 | 0 | 0
Completed | 26 | 23 | 0 | 0
Not Completed | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Period: Second Intervention (Week 24 to Week 72)
Arm/Group | Placebo | Ustekinumab | Placebo to Ustekinumab | Ustekinumab Through End of Study (EOS)
Started | 0 | 0 | 26 | 23
Completed | 0 | 0 | 24 | 23
Not Completed | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ustekinumab | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (13.41) | 54.2 (11.62) | 54.4 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 10 | 5 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 26 | 25 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  JAPAN | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Minimal Improvement in International Myositis Assessment and Clinical Studies Total Improvement Score (IMACS TIS) at Week 24
Description: Minimal improvement was defined as IMACS TIS greater than or equal to (>=) 20 in participants with polymyositis (PM)/dermatomyositis (DM). Criteria used the 6 IMACS core set measures: physician global activity (PhGA)(0-10), patient global activity (PtGA)(0-10), manual muscle testing-8 (MMT-8)(0-80), muscle enzymes (creatine kinase, Aldolase, lactate dehydrogenase, aspartate aminotransferase, alanine aminotransferase), extramuscular assessment of myositis disease activity assessment tool (MDAAT)(0-10), and health assessment questionnaire disability index (HAQ-DI)(0-3). Absolute percent change in each core set measure was calculated as final value minus baseline value divided by range*100. Total improvement score was calculated by sum of 6 core set improvement scores. Total improvement score ranged from 0 to 100 where higher scores indicated greater improvement. This was categorized into 3 categories (minimal [improvement >=20], moderate [improvement >=40] and major [improvement >=60]).
Time Frame: Week 24
Population: All randomized analysis set included all participants who were randomized in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab
Number analyzed (Participants) | 26 | 25
Percentage of participants | 61.5 | 64.0

2. Secondary Outcome: Change From Baseline in Functional Index-2 (FI-2) at Week 24
Description: Change from baseline in FI-2 at Week 24 was reported. The FI-2 was a functional outcome developed for participants with adult PM or DM to assess muscle endurance in 7 muscle groups (shoulder flexion [0-60], shoulder abduction [0-60], head lift [0-60], hip flexion [0-60], step test [0-60], heel lift [0-120], and toe lift [0-120]). Each muscle group was scored as the number of correctly performed repetitions with 60 or 120 maximal number of repetitions depending on muscle group. The FI-2 was performed unilaterally, preferably on the participant's dominant side for muscle groups of shoulder, hip, and step test. The FI-2 score ranged from 0-60 or 0-120 depending on the muscle group. Higher score indicated better muscle endurance.
Time Frame: Baseline, Week 24
Population: All randomized analysis set included all participants who were randomized in this study. Here, 'n' (number analyzed) signifies participants who were evaluable for this outcome measure for given categories.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ustekinumab
Number analyzed (Participants) | 26 | 25
Scores on a scale
  Change in Shoulder Flexion | 2.92 (14.672) | 6.88 (14.284)
  Change in Head Lift | 2.00 (11.331) | 5.56 (13.364)
  Change in Hip Flexion | 2.54 (6.819) | 5.84 (13.184)
  Change in Step Test | 4.15 (10.806) | 3.76 (16.674)
  Change in Heel Lift: number analyzed (Participants) | 26 | 24
  Change in Heel Lift | 1.27 (20.232) | 5.38 (29.315)
  Change in Toe Lift | -0.62 (17.422) | 10.60 (33.800)
  Change in Shoulder abduction | -0.69 (11.589) | 9.00 (15.419)

3. Secondary Outcome: Percentage of Participants Who Experienced Disease Worsening Up to Week 24 Based on Consensus Criteria for Worsening
Description: Percentage of participants who experienced disease worsening up to Week 24 based on consensus criteria for worsening was reported. Criteria for disease worsening in a clinical trial were based on international consensus guideline developed by the IMACS. The worsening of disease was defined as 1 of the following criteria: Worsening of the Physician Global Activity by >=2 centimeter (cm) on a 10-cm visual analogue scale (VAS) and worsening of findings of MMT-8 by >= 20 percent (%) from baseline; worsening of MDAAT-global extramuscular organ disease activity (a composite of constitutional, cutaneous, skeletal, gastrointestinal, pulmonary, and cardiac activity) by >=2 cm on a 10-cm VAS from baseline; worsening of any 3 of 6 IMACS core set (PhGA, PtGA, MMT-8, muscle enzymes, MDAAT, and HAQ-D) activity measures by >= 30% from baseline.
Time Frame: Up to Week 24
Population: All randomized analysis set included all participants who were randomized in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab
Number analyzed (Participants) | 26 | 25
Percentage of participants | 38.5 | 28.0

4. Secondary Outcome: Change From Baseline in Manual Muscle Testing (MMT)-8 Score at Week 24
Description: Change from baseline in MMT-8 score at Week 24 was reported. Manual Muscle Testing was a partially validated tool to assess muscle strength. MMT-8 total score ranged from 0-80, where maximal score was sum of scores from 8 muscle groups (Deltoid middle [left/right], Biceps brachii [left/right], Gluteus maximus [left/right], Gluteus medius [left/right], Quadriceps [left/right], Wrist extensors [left/right], Ankle dorsiflexors [left/right], Neck flexors [axial]) and each muscle group was scored on a 0 to 10-point scale. The sides (right or left) used for calculating the total score. Higher score indicated greater muscle strength, that is, less impairment of muscle.
Time Frame: Baseline, Week 24
Population: All randomized analysis set included all participants who were randomized in this study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ustekinumab
Number analyzed (Participants) | 26 | 25
Scores on a scale | 5.27 (5.647) | 5.88 (5.207)

5. Secondary Outcome: Change From Baseline in Physician Global Activity (PhGA) at Week 24
Description: Change from baseline in PhGA at Week 24 was reported. Physician Global Activity was a partially validated tool to measure the global evaluation by the physician of the participant's overall disease activity at the time of assessment using a 0-10 cm VAS, where 0 cm= no evidence of disease activity and 10 cm= extremely active or severe disease activity. Negative values indicated improvement from baseline.
Time Frame: Baseline, Week 24
Population: All randomized analysis set included all participants who were randomized in this study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ustekinumab
Number analyzed (Participants) | 26 | 25
Scores on a scale | -1.15 (1.623) | -1.22 (2.193)

6. Secondary Outcome: Change From Baseline in Extramuscular Assessment by Myositis Disease Activity Assessment Tool (MDAAT) at Week 24
Description: Change from baseline in extramuscular assessment by MDAAT at Week 24 was reported. This validated tool measure the degree of disease activity of extramuscular organ systems and muscle on a 0-10 cm VAS. Extramuscular activity ranged between 0 and 10 via VAS where, 0 cm = absent and 10 cm = maximum disease activity.
Time Frame: Baseline, Week 24
Population: All randomized analysis set included all participants who were randomized in this study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ustekinumab
Number analyzed (Participants) | 26 | 25
Scores on a scale | -0.68 (1.645) | -1.02 (1.437)

7. Secondary Outcome: Change From Baseline in Muscle Enzyme Levels at Week 24
Description: Change from baseline in muscle enzyme levels (creatine kinase, lactate dehydrogenase) at Week 24 was reported.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Enzyme units per liter (Enzyme U/L)
Arm/Group | Placebo | Ustekinumab
Number analyzed (Participants) | 26 | 25
Enzyme units per liter (Enzyme U/L)
  Creatine Kinase | 140.42 (365.562) | 134.80 (498.102)
  Lactate Dehydrogenase: number analyzed (Participants) | 26 | 24
  Lactate Dehydrogenase | -10.77 (68.577) | -0.67 (64.513)

ADVERSE EVENTS:
Time Frame: Up to Week 88
Description: The safety analysis set included all randomized participants who received at least 1 dose (partial or complete, intravenously [IV] or subcutaneously [SC]) of study agent.
Arm/Group | Placebo | Placebo to Ustekinumab | Ustekinumab Through End of Study (EOS)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/26 | 6/26 | 8/25
Other Adverse Events (participants affected / at risk) | 16/26 | 15/26 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | Placebo to Ustekinumab (N=26) | Ustekinumab Through End of Study (EOS) (N=25)
Glaucoma (Eye disorders) | 0 | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 1
Pneumatosis Intestinalis (Gastrointestinal disorders) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0 | 2
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Cerebral Infarction (Nervous system disorders) | 0 | 2 | 0
Neuroleptic Malignant Syndrome (Nervous system disorders) | 0 | 1 | 0
Anxiety Disorder (Psychiatric disorders) | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | Placebo to Ustekinumab (N=26) | Ustekinumab Through End of Study (EOS) (N=25)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 2
Vitreous Floaters (Eye disorders) | 0 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 2
Oedema Peripheral (General disorders) | 1 | 0 | 2
Vaccination Site Reaction (General disorders) | 2 | 1 | 2
Cellulitis (Infections and infestations) | 2 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4 | 4
Sinusitis (Infections and infestations) | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 2 | 0
Lymphocyte Count Decreased (Investigations) | 2 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Headache (Nervous system disorders) | 2 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 4 | 0 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
This study was terminated early due to lack of efficacy found at Week 24.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT03981744/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT03981744/SAP_001.pdf